CLINICAL TRIAL: NCT00987623
Title: Clinical Evaluation of Two Daily Disposable Lenses in Neophytes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-337-C-031
Record Dates: First submitted 2009-09-29; First posted 2009-10-01 (Estimated); Results first posted 2011-01-13 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nelfilcon A (Experimental): Commercially marketed contact lens worn in both eyes on a daily wear, daily disposable basis for one week.
  Interventions: Device: nelfilcon A contact lens
- narafilcon A (Active Comparator): Commercially marketed contact lens worn in both eyes on a daily wear, daily disposable basis for one week.
  Interventions: Device: narafilcon A contact lens

INTERVENTIONS:
Device: nelfilcon A contact lens — Commercially marketed, hydrogel, single-vision contact lens for daily wear, daily disposable use.
  Arms: nelfilcon A
Device: narafilcon A contact lens — Commercially marketed, silicone hydrogel, single-vision contact lens for daily wear, daily disposable use.
  Arms: narafilcon A

SUMMARY:
The purpose of this study is to evaluate the performance of two daily disposable contact lenses in a population of neophytes (new wearers).

ELIGIBILITY:
Inclusion Criteria:

* No previous contact lens experience or attempts to try contact lenses (neophytes).
* Currently wearing spectacles or needing vision correction in both eyes.
* No older than 45 years of age.
* Able to achieve visual acuity of at least 20/40 in each eye with study lenses in the available parameters.
* Interested in wearing contact lenses.
* Willing to wear study lenses for at least 8 hours/day, at least 5 days/week.
* Other protocol-defined inclusion/exclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks prior to enrollment.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Previous corneal or refractive surgery.
* Currently enrolled in any Clinical Trial.
* Other protocol-defined inclusion/exclusion criteria may apply.

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 326 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Research Intelligence Group (TRiG), Fort Washington, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-seven participants were enrolled but not dispensed. These participants were included in the Actual Enrollment calculation, but not in Participant Flow or Baseline Characteristics calculations.
Period: Overall Study
Arm/Group | Nelfilcon A | Narafilcon A
Started | 145 | 154
Completed | 140 | 151
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Time/job conflict | 2 | 0
Not completed — Discomfort | 1 | 0
Not completed — Biomicroscopy | 0 | 1
Not completed — Influenza | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nelfilcon A | Narafilcon A | Total
Number analyzed (Participants) | 145 | 154 | 299
Age Continuous [Mean (Standard Deviation); unit: years] | 26.5 (9.8) | 26.5 (10.5) | 26.5 (10.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 99 | 193
  Male | 51 | 55 | 106

OUTCOME MEASURES:

1. Primary Outcome: Overall Lens Satisfaction
Description: Overall Lens Satisfaction, as interpreted by the participant and reported on a questionnaire as a single, retrospective evaluation of 1-week's wear time. Overall lens satisfaction was measured on a 10-point scale, with 1 being Poor and 10 being Excellent
Time Frame: 1 week
Population: Analysis conducted per protocol, with exclusions due to major protocol deviations as determined by masked review, discontinuations, and/or missing responses.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Nelfilcon A | Narafilcon A
Number analyzed (Participants) | 128 | 138
Units on a Scale | 7.9 (1.7) | 7.9 (1.6)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the trial: 108 days.
Description: This reporting group includes all enrolled and exposed participants.
Arm/Group | Nelfilcon A | Narafilcon A
Serious Adverse Events (participants affected / at risk) | 0/151 | 0/163
Other Adverse Events (participants affected / at risk) | 0/151 | 0/163

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.